CLINICAL TRIAL: NCT02157038
Title: Neuromuscular Mechanisms Underlying Poor Recovery From Whiplash Injuries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, James Elliott, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00090769
Record Dates: First submitted 2014-05-30; First posted 2014-06-05 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Whiplash Associated Disorders; WAD; Whiplash
Keywords: whiplash; neck pain; chronic pain; motor vehicle accident; car accident; MRI; DNA; RNA
MeSH Terms: conditions — Whiplash Injuries; Neck Pain; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Procedures (Experimental): RNA/DNA blood sample will be collected. Participant will complete questionnaires, MRI and strength and reflex testing.
  Interventions: Device: Pedometer; Device: MRI

INTERVENTIONS:
Device: Pedometer
Device: MRI

SUMMARY:
This study is investigating whether changes in the shape and size of bodily muscles and spinal cord anatomy can influence recovery rates following a motor vehicle collision (MVC). The objective is to demonstrate that the presence of muscle and spinal cord degeneration and associated muscle weakness is the consequence of a mild MVC-related injury involving the cervical spinal cord.

DETAILED DESCRIPTION:
Whiplash is a condition that consists of patients that display varying degrees of pain and disability. Most patients should expect full-recovery within the first 2-3 months post injury. At the other end of the spectrum is a group of patients (~ 25%) who continue to have moderate-severe pain-related disability in the long-term. Reasons for this transition to chronicity are largely unknown. The situation would benefit if there were radiological findings of the disorder. However, clear and consistent findings of injured tissues on standard radiological exams remain elusive.

As part of this study, the investigators will innovatively investigate measures to 1) quantify the temporal development of widespread muscle degeneration, 2) identify quantifiable markers of altered cervical spinal cord physiology, 3) quantify reductions in central activation and fatigue 4) evaluate potential genetic variants that may be associated with chronic pain after a MVC and 5) determine the mediational influence of psychosocial factors on recovery rates following whiplash injury, as a potential mechanism underlying the transition to chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females (18 - 65 years of age)
* Individuals less than one week post MVA with a primary complaint of neck pain.
* Able to give written informed consent and complete interviews in English

Exclusion Criteria:

* Individuals with a spinal fracture from the MVA, or spinal surgeries
* History of one or more MVAs or previous diagnosis of cervical or lumbar radiculopathy
* History of neurological disorders (e.g. Multiple Sclerosis, previous stroke, myelopathy), inflammatory diseases (e.g. Hepatitis, Systemic Lupus Erythematosus, Rheumatoid Arthritis or Osteoarthritis, Alzheimers, Ankylosing Spondylitis, Crohn's disease, Fibromyalgia) or metabolic disorders (e.g. Diabetes, hyper- and hypo-thyroidism)
* Standard contraindications to MRI: claustrophobia, metallic implants, pacemaker and pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2014-07; Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
MRI to assess the changes in markers of altered cervical spinal cord physiology and muscle degeneration. | < 1 week; 2 weeks; 3 months; 1 year of MVC

SECONDARY OUTCOMES:
Neck Disability Index (NDI) Questionnaire | <1 week; 2 weeks, 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors on recovery rates over a period of time.
Coping Strategy Questionnaire-C | < 1 week; 2 weeks; 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Pain Management Inventory (PMI) Questionnaire | < 1 week; 2 weeks; 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Tampa Questionnaire | < 1 week; 2 weeks, 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Post-traumatic Diagnostic Scale (PDS) Questionnaire | < 1 week; 2 weeks; 3 months; 1 year of MVC
  This questionnaire will access the influence and psychosocial factors and recovery rates over a period of time.
Impact of Events Scale Questionnaire | < 1 week; 2 weeks; 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Center for Epidemiological Studies - Depression Scale Questionnaire | < 1 week; 2 weeks; 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Hospital Anxiety and Depression Scale Questionnaire | < 1 week; 2 weeks; 3 months; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Traumatic Injuries Distress Scale and a Symptom Index | < 1 week; 2 weeks; 3 months; 1 year after MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Prediction of Post-MVC Chronic Axial Pain Assessment | Baseline visit
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Follow-Up Data Collection Form for clinical prediction | 2 week; 3 month; 1 year of MVC
  This questionnaire will access the influence of psychosocial factors and recovery rates over a period of time.
Pedometer: wear for 2 consecutive weeks | 2 weeks; 3 months after MVC
  The pedometer will record changes in activity level.
RNA and DNA blood collection | within a week of MVC
  The samples will evaluate potential genetic variants that may be associated with chronic pain after a MVC.
Strength and reflex testing in the lower leg | 2 weeks; 3 months; 1 year
  This testing will demonstrate changes in central activation and fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: James M Elliott, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Smith AC, Laguna JM, Wesselink EO, Scott ZE, Jenkins H, Thornton WA, Wasielewski M, Connor J, Delp S, Chaudhari AS, Parrish TB, Mackey S, Elliott JM, Weber KA 2nd. Leg Muscle Volume, Intramuscular Fat and Force Generation: Insights From a Computer-Vision Model and Fat-Water MRI. J Cachexia Sarcopenia Muscle. 2025 Feb;16(1):e13735. doi: 10.1002/jcsm.13735. PMID 39972963
- [Derived] Callan B, Walton DM, Cleland J, Kolber MJ, Elliott JM. Exploring sex as a moderator of other prognostic variables in whiplash associated disorder: An observational study. PLoS One. 2023 Apr 26;18(4):e0282640. doi: 10.1371/journal.pone.0282640. eCollection 2023. PMID 37099498
- [Derived] Elliott JM, Walton DM, Albin SR, Courtney DM, Siegmund GP, Carroll LJ, Weber KA 2nd, Smith AC. Biopsychosocial sequelae and recovery trajectories from whiplash injury following a motor vehicle collision. Spine J. 2023 Jul;23(7):1028-1036. doi: 10.1016/j.spinee.2023.03.005. Epub 2023 Mar 21. PMID 36958668
- [Derived] Modarresi S, MacDermid JC, Suh N, Elliott JM, Walton DM. How Is the Probability of Reporting Various Levels of Pain 12 Months After Noncatastrophic Injuries Associated with the Level of Peritraumatic Distress? Clin Orthop Relat Res. 2022 Feb 1;480(2):226-234. doi: 10.1097/CORR.0000000000002024. PMID 34705736